CLINICAL TRIAL: NCT06094764
Title: Measuring the Effectiveness of a Personal Cooling Vest for the Prevention of Heat Strain in Construction Workers
Brief Title: S&B Heat Stress Pilot Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, William B Perkison, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-22-0651
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Thermal Discomfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Personal monitoring device and a cooling vest , Then personal monitoring device only (Experimental)
  Interventions: Device: Group A
- Personal monitoring device only, Then personal monitoring device and a cooling vest (Experimental)
  Interventions: Device: Group B

INTERVENTIONS:
Device: Group A — The intervention will take place after lunch for about 2-3 hours in regular working conditions. Group A will be fitted with a cooling and bio-harness. At the end of each workday, participants will return the monitors and vests will be removed and returned to the research station. The biomonitor's battery will be recharged and data downloaded. The ice vests will be placed in a freezer.
  Arms: Personal monitoring device and a cooling vest , Then personal monitoring device only
Device: Group B — The intervention will take place after lunch for about 2-3 hours in regular working conditions. Group B will wear a bio-harness and no cooling vest.At the end of each workday, participants will return the monitors and vests will be removed and returned to the research station. The biomonitor's battery will be recharged and data downloaded. The ice vests will be placed in a freezer.
  Arms: Personal monitoring device only, Then personal monitoring device and a cooling vest

SUMMARY:
The purpose of this study is to develop a heat stress program for the construction industry and evaluate its feasibility and appeal.

ELIGIBILITY:
Inclusion Criteria:

* employed at S&B
* work more than 20 hours a week

Exclusion Criteria:

* severe chronic disease (e.g. severe pulmonary or cardiovascular disease
* history of severe heat stroke
* use of a pacemaker
* any medical issue which would render the participant unable to wear a chest monitor and cooling vest.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Thermal discomfort as assessed by the thermal comfort scale | end of study (about 2 hours after start)
  The thermal comfort scale is a 7-point scale that asks participants to rate their level of thermal comfort ranging from the sensation of "cold, cool, slightly cool, neutral, slightly warm, warm, hot

SECONDARY OUTCOMES:
Change in Heart rate as assessed by the Zephyr BioHarness 3.0 device | from baseline to end of study (2 hours after baseline)
Estimated core body temperature as assessed by the Zephyr BioHarness 3.0 device | from baseline to end of study (2 hours after baseline)
Respiratory rate as assessed by the Zephyr BioHarness 3.0 device | from baseline to end of study (2 hours after baseline)
Caloric burn as assessed by the Zephyr BioHarness 3.0 device | from baseline to end of study (2 hours after baseline)
Hydration status as indicated by urine specific gravity as assessed by a clinical refractometer analysis of urine sample | from baseline to end of study (2 hours after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: William Perkison, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No